CLINICAL TRIAL: NCT06582199
Title: Precision Medicine in Alzheimer's Disease: Integration of Resilience Metrics and Risk Factors - Validation Cohort BioCogBank-AD
Brief Title: Precision Medicine in Alzheimer's Disease : Integration of Resilience Metrics and Risk Factors - Validation Cohort BioCogBank-AD
Acronym: BioCogBank-AD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: National Research Agency, France (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Centre National de la Recherche Scientifique, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: APHP210991; 2024-A00457-40 (Other: ID-RCB)
Record Dates: First submitted 2024-07-23; First posted 2024-09-03 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-12

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer Disease; Mild cognitive impairment; Resilience; Biomarkers; Cohort; Clinical practice
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Exploratory group (Experimental)
  Interventions: Other: Blood sample; Behavioral: Neuropsychological battery tests

INTERVENTIONS:
Other: Blood sample — Plasma, DNA, RNA and PBMC Sampling
Behavioral: Neuropsychological battery tests — * Short term memory: Digit span (forward and backward)
  * Long term memory: Free and Cued selective reminding Test
  * Language and semantic Memory : Verbal Fluency (Category and Litteral), Image Naming (DO 40)
  * Praxis
  * Visuo Spatial abilities: Rey-Osterrieth Complex Figure Test
  * Attention and executive functions: Trail Making Test (TMT) Part A and B, Frontal Assessment Battery (FAB)
  * Autonomy in daily life activities : Alzheimer's Disease Cooperative Study - Activities of Daily Living Inventory (ADCS-ADL), Instrumental Activities of Daily Living (IADL)
  * Mood and anxiety: Hospital Anxiety and Depression Scale (HADS)
  * Cognitive reserve : Cognitive Reserve Index questionnaire (CRIq)

SUMMARY:
BioCogBankAD aims at building a prospective clinical practice cohort of 244 patients with biologically confirmed mild cognitive impairment due to Alzheimer's Disease (AD) or mild AD in order to validate data regarding markers of resilience toward AD pathophysiological process discovered in an upstream project called AD-Resilience.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is a leading cause for individual and caregiver burden associated with neurodegenerative diseases (NDs) in an aging population, afflicting + 35 million people worldwide, and spiraling costs. Major advances have been made during the last 20 years in the understanding of AD pathophysiological process. It is now well demonstrated that the course of the disease extend over more than 20 years with long pre and pauci-symptomatic periods.

A major need and challenge in translational research on Alzheimer's disease (AD) is to predict disease progression rate and/or time to clinical conversion, notably in the early phases of the AD process, such as mild cognitive impairment (MCI). Current markers such as Aß and tau species measured in cerebrospinal fluid (CSF) can differentiate AD from control and are currently used in daily clinical practice to assess presence of AD pathological process in patients with cognitive complaints. However, they do not account for cellular compensation and resistance mechanisms, the so-called "resilience" process.

Consequently, both prediction of AD progression in single patients and personalized adaptation of management and treatment remain highly limited. Moreover, there is an important unmet need regarding targeted prevention.

AD-Resilience is a translational research study funded by Agence Nationale pour la Recherche (ANR) and Direction Générale de l'Organisation des Soins (DGOS) that aims at identifying and validating markers of the biological processes underlying the mechanisms of brain resilience toward AD pathological process. Using blood samples, the investigators will produce the molecular-profile data that are needed to assess the resilience and brain homeostasis status of patients facing the AD process. Results will be processed using high-end machine learning (ML) to overcome the limitations associated with sub-optimal reliability and precision of dimensional data analysis.

These biomarkers will be identified using data and samples from an already available nationwide research cohort (BALTAZAR). In order to ensure validity and facilitate transfer to clinical practice, results from this preliminary study will have to be confirmed in an independent, prospective cohort of patients reflecting the full spectrum and real-life heterogeneity of AD.

For this purpose, BioCogBankAD study aims at building this validation cohort. 244 patients with MCI or early dementia due to AD will be recruited in the present study and prospectively followed during three years. Blood samples (plasma, DNA and PaxGen) will be taken from these patients in order to measure the biomarkers previously identified in the exploratory study. Clinical follow-up including including standardized neuropsychological examination and blood sampling (plasma) will be performed annually.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AD according to IWG-2 2014 criteria
* Age 50-90 year old
* Affiliated or beneficiary of a social security scheme
* MMSE ≥ 20
* Abnormal CSF Aβ42 or Aβ40/Aβ42 ratio according to local cut-offs
* Abnormal CSF phosphorylated and total Tau according to local cut-offs
* Ability to pass neuropsychological assessments
* Availability of a brain MRI with T1 volumetric sequence performed within 1 year

Exclusion Criteria:

* Other cause of dementia
* Participation in an AD therapeutic clinical trial
* Protected adults (including individual under guardianship by court order),

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Mean levels of new blood biomarkers | 36 months
  assess biomarkers of biological resilience toward AD pathological process

SECONDARY OUTCOMES:
Mini-Mental State examination (MMSE) | 36 months
  assess relationship between new biomarkers (biomarkers identified in the current study on the analysis of study samples Baltazar) and cognitive decline - MMSE: 0 to 30 evaluates memory, orientation in space and time, learning and immediate memory, attention and reasoning, language and ability to perform tasks.
  * Score of 27 or more: no cognitive impairment
  * Score between 21 and 26: slight impairment
  * Score between 11 and 20: moderate impairment
  * Score below 10: severe impairment
Cognitive performance (zScore) | 36 months
  assess relationship between new biomarkers (biomarkers identified in the current study on the analysis of study samples Baltazar) and cognitive decline -
Instrumental Activities of Daily Living (IADL) | 36 months
  assess relationship between new biomarkers and loss of autonomy (decline on IADL) - 0 dependent to 17 Assessment of autonomy in instrumental activities of daily living - The score shows the level of autonomy: a maximum score represents maximum autonomy, and the lower the score, the lower the level of autonomy.
Hospital Anxiety and Depression Scale (HADS) | 36 months
  The HAD scale is a screening instrument for anxiety and depressive disorders. It comprises 14 items rated from 0 to 3. Seven questions relate to anxiety (total A) and seven to depression (total D), giving two scores (maximum score for each = 21).
  0 = no anxiety 21= anxiety and depressive disorders max
Cognitive Reserve Index questionnaire (CRIq) | 36 months
  CRI schooling min = 0 no schooling, training or internship - Max = undefined because "+1" corresponds to each year of schooling and +0.5 for any internship of more than 6 months - CRI work is the number of years of work, rounded to a scale of 5 (0-5-10-15-20) to assess the degree of intellectual effort and personal responsibility - CRI leisure from never/rarely to often/always (checkboxes) multiplied by number of years of practice.
  Score CRI :
  * ≤70 = low
  * 70 to 84 = low average
  * 85 to 114 = average From 115 to 130 = high average
  * ≥ = high
Cerebrospinal Fluid (CSF) biomarkers of AD | 36 months
  correlate the new blood biomarkers levels and CSF biomarkers of AD (Aβamyloid, Tau, P Tau)

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel GOGNAT, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris; Christian NERRI, PhD, Study Chair — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Hôpital Cochin, Paris, France

IPD SHARING:
Plan to Share IPD: No